CLINICAL TRIAL: NCT00388947
Title: The Prolapse Registry: An Observational Collection of Short- and Long-Term Patient Outcomes Following Use of AMS Surgical Devices for the Repair of Female Genital Prolapse
Brief Title: Observational Data Collection of Surgical Outcomes in the Treatment of Vaginal Prolapse With AMS Products
Acronym: POWER1012
Status: Completed | Type: Observational
Sponsor: ASTORA Women's Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 1012
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Vaginal Prolapse
Keywords: vaginal prolapse; cystocele; rectocele; enterocele; apical prolapse; vaginal vault prolapse
MeSH Terms: conditions — Uterine Prolapse; Cystocele; Rectocele; Hernia; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: AMS Prolapse Product (AMS Apogee™ with IntePro (Synthetic) or InteXen (Biologic) Mesh implant for posterior wall pelvic organ prolapse AMS Straight-In™ with IntePro (Synthetic) Mesh implant for vaginal vault pelvic organ prolapse AMS Perigee™ with IntePro Mesh implant for anterior wall pelvic organ prolapse AMS Perigee™ with IntePro Mesh coated with PC AMS Elevate® Prolapse Repair System Family)
  Interventions: Device: AMS Prolapse Product

INTERVENTIONS:
Device: AMS Prolapse Product — AMS Apogee™ with IntePro (Synthetic) or InteXen (Biologic) Mesh implant for posterior wall pelvic organ prolapse AMS Straight-In™ with IntePro (Synthetic) Mesh implant for vaginal vault pelvic organ prolapse AMS Perigee™ with IntePro Mesh implant for anterior wall pelvic organ prolapse AMS Perigee™ with IntePro Mesh coated with PC AMS Elevate® Prolapse Repair System Family
  Other Names: Apogee, Straight-In, Perigee, Elevate anterior, Elevate Posterior

SUMMARY:
This registry was observational (only collected information typically noted by the surgeon when their patients were routinely seen); there was no change to the care the patient received as a result of being part of the registry). Data collection focused on the surgical outcomes of AMS prolapse products.

DETAILED DESCRIPTION:
The Prolapse Registry was an observational study of patients who were implanted with AMS devices for the surgical repair of female pelvic prolapse. The registry followed patients post-operatively for up to 2 years and collected demographic, clinical, surgical, safety, and patient outcomes data.

The registry was a web-based system in which surgeons entered patient information with regard to their prolapse surgery. All information entered was de-identified (no names, no date of birth, no date of surgery, etc).

ELIGIBILITY:
Inclusion Criteria:

* Female at least 21 years old
* Has pelvic organ prolapse requiring surgical repair
* Receives at least one of the AMS Prolapse Repair devices in the treatment of their pelvic organ prolapse

Exclusion Criteria:

* Is contraindicated for an AMS Prolapse Repair per the product's Instruction for Use.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects greater than or equal to 21 years of age with genital prolapse who undergo surgical reconstruction of the pelvic floor using an AMS Prolapse Repair device.
Sampling Method: Non-Probability Sample
Enrollment: 1543 (Actual)
Dates: Start 2006-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Zylstra, MD, Principal Investigator — Whitinsville Medical Center
Locations (1):
- Samuel Zylstra, MD, Whitinsville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was registered in September 2006, The last patient data were entered in May 2010.
Pre-assignment Details: Patients had to met all of the inclusion criteria and none of the exclusion criteria.
Groups:
- 1 - Any AMS Prolapse Product: at least one AMS prolapse product was used
Period: Overall Study
Arm/Group | 1 - Any AMS Prolapse Product
Started | 1590
Completed | 1543 (47 patients excluded because no AMS prolapse device was noted.)
Not Completed | 47
Not completed — Protocol Violation | 47

BASELINE CHARACTERISTICS:
Arm/Group | 1 - Any AMS Prolapse Product
Number analyzed (Participants) | 1590
Age, Continuous [Mean (Standard Deviation); unit: participants] — Patients >89 years old were excluded because protected health information was not collected in this study. Mean age excludes patients >89 years old. Two patients were >89 years old.
  participants
    Age <89 years | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1590
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients With at Least One Adverse Event Related to Any AMS Prolapse Device
Time Frame: up to 2-years post-implant
Population: All patients that met the inclusion/exclusion criteria.
Measure: Number; unit: participants
Arm/Group | 1 - Any AMS Prolapse Product
Number analyzed (Participants) | 1543
participants | 194

2. Secondary Outcome: Prolapse Efficacy Success Rate
Description: Success was defined as either (1) Baden-Walker grade 0 or 1 or (2) (Pelvic Organ Prolapse Quantification System) POP-Q stage 0 or 1. If a site reported both measurements, then the POP-Q score was used.
Time Frame: 24 months
Population: Patients returning for a visit between 19-24 months post-procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1 - Any AMS Prolapse Product
Number analyzed (Participants) | 332
percentage of participants | 81.6 [77.0 to 85.6]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 1 - Any AMS Prolapse Product
Serious Adverse Events (participants affected / at risk) | 71/1543
Other Adverse Events (participants affected / at risk) | 138/1543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Any AMS Prolapse Product (N=1543)
Adhesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dehiscence at vaginal suture line before healing occurs (Surgical and medical procedures) | 2 (2)
Extrusion (General disorders) | 24 (26)
Granuloma formation (Skin and subcutaneous tissue disorders) | 2 (2)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Incontinence (Renal and urinary disorders) | 6 (6) — includes denovo and recurrent incontinence
Infection (Infections and infestations) | 1 (1)
Other Genitourinary (General disorders) | 2 (2) — 1)Coumadin medicated patient received too much anticoagulation therapy resulting in bleeding 2)small separation of anterior mesh from vaginal mucosa
Pain - dyspareunia (General disorders) | 2 (2)
Pain - excluding dyspareunia (General disorders) | 3 (3)
Perforation - bladder (Injury, poisoning and procedural complications) | 5 (5)
Prolapse (Reproductive system and breast disorders) | 14 (14) — includes denovo and recurrent
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary urge, frequency, or hesistancy (Renal and urinary disorders) | 2 (2)
Wound separation <3 months post-op (General disorders) | 3 (3) — Wound separation events less than 3 months post-procedure including mesh exposure events
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Any AMS Prolapse Product (N=1543)
extrusion (General disorders) | 30 (32) — mesh exposure through vaginal mucosa
granuloma formation (Skin and subcutaneous tissue disorders) | 11 (11)
hematoma (Surgical and medical procedures) | 10 (10)
incontinence (Renal and urinary disorders) | 12 (12) — Includes both denovo and worsening incontinence
infection (Infections and infestations) | 13 (14)
other events below threshold (Skin and subcutaneous tissue disorders) | 28 (28) — Incongruous events that are individually below the threshold
pain (excluding dyspareunia) (General disorders) | 15 (15)
prolapse (Reproductive system and breast disorders) | 40 (41) — includes denovo and recurrent prolapse

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AMS (sponsor) is the sole owner of the conglomerate data inputted into the POWER database and has the right to publish such data at its sole discretion. Registry Physician will provide AMS with a copy of any data, finding, result, article, abstract, manuscripts, presentation, or other information intended for publication, at least thirty (30) days prior to submission of same for publication.